CLINICAL TRIAL: NCT06251362
Title: The Impact of Sleep Restriction on Physical Performance, Markers of Muscle Damage, Inflammation, and Brain-derived Neurotrophic Factor (BDNF) Levels in Female Soccer Players.
Brief Title: Effects of Sleep Restriction on Female Soccer Players: Physical Performance, Muscle Damage, Inflammation, and BDNF Levels.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Collaborators: Jagiellonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: SKN/SP/570683/2023
Record Dates: First submitted 2023-12-12; First posted 2024-02-09 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-02

CONDITIONS: Sleep; Sleep Restriction
Keywords: acute sleep restriction; early sleep restriction; female athletes; football

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sleep (No Intervention): The night before the experimental session, where participants will follow their habitual sleep-wake routines.
- Sleep restriction (Experimental): The night before the experimental session (with sleep restrictions (SR)), where participants will experience acute sleep restriction the night before the test session (i.e., 3 h of early sleep restriction versus normal sleep).
  Interventions: Procedure: Sleep restriction

INTERVENTIONS:
Procedure: Sleep restriction — Participants will experience a night of acute sleep restriction. During this night, they will sleep 3 hours less than usual.
  Arms: Sleep restriction

SUMMARY:
This research aims to investigate the interplay between menstrual cycles, sleep patterns, and athletic performance. Before experimental sessions, participants will maintain menstrual diaries for three months and complete assessments for sleep disorders and chronotype. Sleep duration will be objectively measured over five nights using actigraphy, complemented by sleep-related data from an actigraph and the Karolinska Sleep Diary.

The study involves two sessions: normal sleep (based on habitual duration) and restricted sleep (reduced by 3 hours). Athletes will engage in a simulated match-play game before both sessions, followed by comprehensive performance tests the next day. Blood samples will be collected at three intervals to analyze hormonal profiles (including progesterone, and estradiol), markers of muscle damage, inflammation, stress (such as TNF-α, IL-6, CRP, myoglobin, cortisol, testosterone), and brain-derived neurotrophic factor (BDNF).

On Day 1, pre- and post-training blood samples will be obtained, and participants will wear an actigraph, adhere to specified bedtime routines, and report activities (restricted sleep group). Day 2 involves completing a sleep diary, refraining from caffeine, responding to questionnaires assessing readiness to train and mood, and undergoing performance tests followed by self-reporting of pain levels and perceived exertion using established scales (VAS, RPE 6-20).

DETAILED DESCRIPTION:
Before commencing experimental sessions, the menstrual cycles of the participants will be assessed using a menstrual diary spanning three months before the sessions. Additionally, each athlete will be asked to complete a questionnaire for screening sleep disorders (PSQI) and a chronotype classification questionnaire (MEQ). The average sleep duration over five consecutive nights will be measured using actigraphy; this analysis will determine the length of sleep allocated during experimental sessions. Sleep-related parameters will be recorded using an actigraph (MotionWatch8) and confirmed using the Karolinska Sleep Diary (KSD).

The project involves two experimental sessions (each spanning two days) under two different conditions: a) normal sleep (NS; habitual sleep duration determined from the analysis of five consecutive nights) and b) restricted sleep (RS; sleep reduced by 3 hours during the nocturnal period compared to NS). Participants will perform a simulation match-play game (SAFT90) before NS and RS, followed by performance tests on the following day. Blood samples will be collected at three-time points: a) pre-training, b) post-training, and c) before morning tests on the second day of the experiment. Biochemical analysis of the blood will include progesterone and estradiol (for menstrual cycle analysis) as well as parameters related to muscle damage, inflammatory state, and stress levels (TNF-α; IL-6; CRP; myoglobin; hematology; cortisol; testosterone). Additionally, the level of brain-derived neurotrophic factor (BDNF) will be analyzed.

Day 1 of the experiment: Immediately before training, the first blood collection (8 ml) will occur to analyze the necessary blood biochemical parameters. Subsequently, athletes will undergo a standardized afternoon training session, including a simulation match-play game (SAFT90). Another blood sample will be taken immediately after the exercise. Participants will be asked to wear an actigraph on their non-dominant wrist and consume dinner according to the provided recommendations. They will be instructed to go to bed according to a specified schedule (NS or RS). Additionally, participants will be instructed to spend the time before bedtime engaged in routine evening activities (excluding stimulants like coffee or additional exercise). Participants with restricted sleep will also be requested to report their activities every 30 minutes until they go to bed using an internet communicator.

Day 2 of the experiment: Participants will complete the Karolinska Sleep Diary upon waking up. They will also be asked to abstain from consuming caffeine-containing foods and to have breakfast following the provided recommendations. Before the session begins, participants will complete a readiness to train questionnaire (RTQ) and a mood assessment questionnaire (POMS). Blood samples will be collected, followed by specific football-related performance tests: a) repeated high-intensity effort capacity (Yo-Yo test); b) lower limb power (vertical jump); c) maximal acceleration (3x30 m sprints); d) agility with and without the ball (Zig-Zag Test). Immediately after the performance tests, participants will indicate their pain level (Visual Analogue Scale; VAS) and rate their perceived exertion (RPE 6-20).

ELIGIBILITY:
Inclusion Criteria:

* a minimum of 5 years of training experience
* practicing physical activity for the last 6 months at least 3 times per week for 2h
* current medical qualification for competitive sport

Exclusion Criteria:

* diseases that can have a bad influence on the menstrual cycle (e.g. polycystic ovarian syndrome, endometriosis);
* using hormonal contraception;
* regularity of the menstrual cycle.
* diagnosed cardiovascular, metabolic, gastrointestinal, or neurological diseases; movement, neuromuscular or musculoskeletal disorders;
* taking medications and supplements that may affect fitness test results; taking supplements that may affect biochemical test results
* sleep disorders (PSQI >5)

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Countermovement jump | 1 day after night with or without intervention
  Vertical jump test performed by having an athlete quickly squat to a self-selected depth and then jump as high as possible.
Sprint test (0-30m) | 1 day after night with or without intervention
Zig Zag test | 1 day after night with or without intervention
Zig Zag test with ball | 1 day after night with or without intervention
Yo-Yo Intermittent endurance test level I | 1 day after night with or without intervention
Flanker task | 1 day after night with or without intervention

SECONDARY OUTCOMES:
Mood (POMS) | 1 day after night with or without intervention. During each experimental session. Before sports performance protocol
  The POMS is a widely-applied measure for the assessment of an individual's mood.
Pain (Pain scale) | 1 day after night with or without intervention. Immediately after the last performance exercise in experimental sessions
  A pain scale is a tool use to help assess a person's pain. Scale 0 (lack of pain) 10 (maximum pain)
Readiness-to-train questionnaire (RTT-Q) | 1 day after night with or without intervention. During each experimental session. Before sports performance protocol
  Subjective reactions related to the level of motivation for effort
Rating perceived exertion (RPE) | 1 day after night with or without intervention. Immediately after the last performance exercise in experimental sessions
  A subjective scale that assesses the severity of effort exerted. Includes a rating from 6 perceiving "no effort" to 20 perceiving "maximum effort."
Stress and recovery (SRSS) | 1 day after night with or without intervention. In the morning, each experimental day and the day after
  The Short Recovery and Stress Scale (SRSS) measure the recovery-stress state of an athlete multidimensionally with eight items on emotional, mental, physical, and overall levels.

OTHER OUTCOMES:
Objective Sleep - Total sleep time | 1 day after night with or without intervention. The night before and after the experimental sessions
  Total sleep time obtained from sleep onset to time at wake-up assessed by actigraphy
Objective Sleep - Sleep efficiency | 1 day after night with or without intervention. The night before and after the experimental sessions
  The percentage of total sleep time to lights off and leaving bed assessed by actigraphy
Objective Sleep - WASO (Wake After Sleep Onset) | 1 day after night with or without intervention. The night before and after the experimental sessions
  The total number of minutes that a person is awake after having initially fallen asleep assessed by actigraphy
Objective Sleep - Sleep duration | 1 day after night with or without intervention. The night before and after the experimental sessions
  The quantity of time that a person sleeps assessed by actigraphy
Objective Sleep - Sleep onset time | 1 day after night with or without intervention. The night before and after the experimental sessions
  The time it takes a person to fall asleep after turning the lights out assessed by actigraphy
Objective Sleep - Wake time | 1 day after night with or without intervention. The night before and after the experimental sessions
  The hours in the day that a person is awake assessed by actigraphy
Blood collection - progesterone | 1 day after night with or without intervention. Before each experimental sesion
  Blood will be drawn to measure progesterone
Blood collection - estradiol | 1 day after night with or without intervention. Before each experimental sesion
  Blood will be drawn to measure estradiol
Blood collection - cortisol | Before and after the match simulation and before the experimental session on the second day 1 day after night with or without intervention.
Blood collection - testosterone | 1 day after night with or without intervention. Before and after the match simulation and before the experimental session on the second day
Blood collection - TNF-α | 1 day after night with or without intervention. Before and after the match simulation and before the experimental session on the second day
Blood collection - IL-6 | 1 day after night with or without intervention. Before and after the match simulation and before the experimental session on the second day
Blood collection - CRP | 1 day after night with or without intervention. Before and after the match simulation and before the experimental session on the second day
Blood collection - myoglobin | 1 day after night with or without intervention. Before and after the match simulation and before the experimental session on the second day
Blood collection - brain-derived neurotrophic factor (BDNF) | 1 day after night with or without intervention. Before and after the match simulation and before the experimental session on the second day
Karolinska Sleep Diary (KSD) | 1 day after night with or without intervention. The morning of the session and the next day after the experimental session

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - The Academy of Physical Education in Krakow, Krakow
  - University School of Physical Education in Cracow, Krakow